CLINICAL TRIAL: NCT06539000
Title: The "RIGHT-SCORE" Study: a Preoperative Risk Score for Postoperative Right Ventricular Dysfunction in Adult Cardiac Surgery
Brief Title: Preoperative Risk Score for Postoperative Right Ventricular Dysfunction in Adult Cardiac Surgery
Acronym: The RightScore
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Principal Investigator, Alessandro Strumia, MD, Dr., Fondazione Policlinico Universitario Campus Bio-Medico
Other Study IDs: The RightScore
Record Dates: First submitted 2024-07-21; First posted 2024-08-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Right Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction, Right

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Right ventricular dysfunction (RVD) is common following cardiac surgery, and it is characterised by impaired right ventricular function that can lead to decreased cardiac output and hemodynamic instability. RVD is consistently associated with poor outcomes.

The mechanisms behind RVD post-surgery involve changes in preload, after load, and RV contraction. Factors linked to higher incidence of postoperative RVD include decreased tricuspid annular plane excursion (TAPSE), elevated preoperative pulmonary artery pressure, lung diseases, duration of extracorporeal circulation, and left valve surgery.

While predictive scores for RVD exist for left ventricular assist device (LVAD) patients, no such models are available for other cardiac surgeries. Identifying specific predictors could lead to models that identify high-risk patients, allowing for tailored monitoring and treatment strategies.

The primary aim of this study is to create a preoperative risk score for predicting the development of right ventricular dysfunction following adult cardiac surgery through a retrospective analysis on patients who underwent heart surgery.

DETAILED DESCRIPTION:
Postoperative RVD will be defined as:

- Echocardiographic parameters suggestive of RVD (at least 2 out of 3): TAPSE < 16 mmHg; right ventricular fractional area change (RVFAC) < 35%; right ventricular end systolic dilation > 3,5 cm (measured from the septum to the free wall).

AND

- Need for inotropic and/or pulmonary vasodilator drug support and/or mechanical support.

Data will be collected retrospectively on: demographic characteristics; basic patient characteristics (weight, height, Body Mass Index -BMI, etc.); preoperative pharmacological therapy; preoperative comorbidities; abnormalities in blood tests; chest X-rays and ECGs; abnormalities in coronary angiography and carotid ultrasound; preoperative echocardiographic examination: TAPSE, Left Ventricular Ejection Fraction- LVEF, valvular pathologies, Pulmonary Artery Systolic Pressure- PAPs, pericardial effusion; type of surgical intervention; occlusion of the posterior interventricular coronary artery (acute or chronic); duration of the surgical procedure; duration of extracorporeal circulation; non-revascularized right coronary artery disease; blood product transfusions; postoperative pharmacological therapy (with particular regard to the use of inotropes/pulmonary vasodilators/vasopressors); postoperative echocardiographic examination: TAPSE; RVFAC; right ventricular dilation at end-systole; postoperative complications; Intensive Care Unit (ICU) length of stay and hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* elective or urgent cardiac surgery at Campus BioMedico between January 2016 to December 2023
* postoperative echocardiogram execution
* ASA class I-IV

Exclusion Criteria:

* age < 18 years
* inotropic therapy at the time of surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent cardiac surgery between January 2016 and December 2023 at the Policlinico Fondazione Campus BioMedico.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Creation of a preoperative risk score for predicting the development of right ventricular dysfunction after adult cardiac surgery. | September 2024 - December 2025
  Preoperative patient characteristics (demographic features, BMI, preoperative conditions, etc.) and surgical factors (type of procedure, duration of cardiopulmonary bypass, duration of surgery, etc.) will be correlated with the development of RVD in the early postoperative period. Scores will be assigned to factors showing significant correlation. The sum of these scores will yield the total score and thus the risk level.
  Unabbreviated score title: The RightScore
  Minimum/maximum values: Depending on the number of risk factors associated with right ventricular dysfunction.
  Higher scores indicate worse outcomes.

SECONDARY OUTCOMES:
Retrospective validation of the created score (The RightScore) on adult cardiac surgery patients operated at Policlinico Fondazione Campus Bio-Medico between January 2016 and December 2023. | September 2024 - December 2025
  The RightScore will be calculated using retrospectively analyzed data for every adult patient operated on at Policlinico Fondazione Campus Bio-Medico between January 2016 and December 2023. Preoperative and intraoperative data will be used to predict postoperative right ventricular dysfunction. This prediction will be correlated with the actual development of postoperative right ventricular dysfunction to retrospectively validate the score created.
  Unabbreviated score title: The RightScore
  Minimum/maximum values: Depending on the number of risk factors associated with right ventricular dysfunction.
  Higher scores indicate worse outcomes.
Correlation between postoperative RVD and postoperative outcomes. | September 2024 - December 2025
  Correlation with mortality, stroke, multi-organ dysfunction, re-intubation, cardiac arrest, increased length of stay in the ICU, increased hospital stay.
Sub-analysis of the risk score. | September 2024 - December 2025
  Sub-analysis of the risk score for the subtype of surgery performed by the patient.
  Unabbreviated score title: The RightScore
  Minimum/maximum values: Depending on the number of risk factors associated with right ventricular dysfunction.
  Higher scores indicate worse outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mattei A, Strumia A, Benedetto M, Nenna A, Schiavoni L, Barbato R, Mastroianni C, Giacinto O, Lusini M, Chello M, Carassiti M. Perioperative Right Ventricular Dysfunction and Abnormalities of the Tricuspid Valve Apparatus in Patients Undergoing Cardiac Surgery. J Clin Med. 2023 Nov 17;12(22):7152. doi: 10.3390/jcm12227152. PMID 38002763
- [Background] Varma PK, Jose RL, Krishna N, Srimurugan B, Valooran GJ, Jayant A. Perioperative right ventricular function and dysfunction in adult cardiac surgery-focused review (part 1-anatomy, pathophysiology, and diagnosis). Indian J Thorac Cardiovasc Surg. 2022 Jan;38(1):45-57. doi: 10.1007/s12055-021-01240-y. Epub 2021 Oct 27. PMID 34898875
- [Background] Estrada VH, Franco DL, Moreno AA, Gambasica JA, Nunez CC. Postoperative Right Ventricular Failure in Cardiac Surgery. Cardiol Res. 2016 Dec;7(6):185-195. doi: 10.14740/cr500e. Epub 2016 Dec 31. PMID 28197291
- [Background] Kaul TK, Fields BL. Postoperative acute refractory right ventricular failure: incidence, pathogenesis, management and prognosis. Cardiovasc Surg. 2000 Jan;8(1):1-9. doi: 10.1016/s0967-2109(99)00089-7. PMID 10661697
- [Background] Matthews JC, Koelling TM, Pagani FD, Aaronson KD. The right ventricular failure risk score a pre-operative tool for assessing the risk of right ventricular failure in left ventricular assist device candidates. J Am Coll Cardiol. 2008 Jun 3;51(22):2163-72. doi: 10.1016/j.jacc.2008.03.009. PMID 18510965

DOCUMENTS (1):
  • Statistical Analysis Plan (2024-07-20): https://cdn.clinicaltrials.gov/large-docs/00/NCT06539000/SAP_000.pdf